CLINICAL TRIAL: NCT01879475
Title: Prospective, Randomised, Controlled Investigation Comparing the Safety and Performance of 032-11 Surgical Haemostat With FLOSEAL® Haemostatic Matrix in Cardiac Surgery and Thoracic Aortic Surgery.
Brief Title: Safety and Performance of 032-11 Haemostat in Cardiac and Thoracic Aortic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medtrade (Industry)
Collaborators: The Clinical Trial Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT001
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: C.Surgical Procedure; Cardiac; Haemorrhage.
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 032-11 (Experimental): 032-11 topical haemostat.
  Interventions: Device: 032-11
- Floseal (R) (Active Comparator): Floseal(R) topical haemostat
  Interventions: Device: Floseal (R)

INTERVENTIONS:
Device: 032-11 — Topical haemostat
  Arms: 032-11
Device: Floseal (R) — Topical haemostat
  Arms: Floseal (R)

SUMMARY:
The effectiveness objective of this study is to evaluate whether 032-11 is non-inferior to Floseal as an adjunct to achieving haemostasis during surgical procedures involving cardiac and aortic thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be equal or greater than 18 years old
* The patient must have elective or non-elective urgent cardiac surgery or thoracic aortic surgery
* The patient must have no childbearing potential or have a negative serum or urine pregnancy test within 7 days of the planned surgery or in the opinion of the Investigator performs adequate contraception
* The patient is willing and able to be contacted for the follow-up visit at 6- 8 weeks
* The patient must provide written informed consent using a form that is reviewed and approved by the IEC

Exclusion Criteria:

* The patient is currently enrolled in this or another investigational device or drug trial that has not completed the required follow up period.
* The patient has a known hypersensitivity to materials of bovine origin
* The patient does not wish to receive materials of bovine or shellfish origin for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Haemostasis success | Intra-operative
  Proportion of patients achieving haemostasis success following the first application of compression.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Millner, MD FRCS, Study Chair — Blackpool Victoria Hospital NHS trust
Locations (1):
- Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire, United Kingdom